CLINICAL TRIAL: NCT03281343
Title: Linkage to Community-Based HIV Pre-Exposure Prophylaxsis Care Among at Risk Women Upon Release From Incarceration
Brief Title: Linking Women to PrEP Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA045621 (NIH)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Prevention
Keywords: PrEP; Women; Linkage to Care
MeSH Terms: interventions — Motivational Interviewing; Patient Navigation; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-NAV (Experimental): A study therapist will deliver a motivational interviewing session with participants while they are incarcerated and serve as a role of patient navigator post-release.
  Interventions: Behavioral: Motivational Interviewing & Patient Navigator
- Standard of Care (SOC) (Active Comparator): Approximates care currently provided at the prison.
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Motivational Interviewing & Patient Navigator — The specific content, structure, and implementation approach for MI-NAV will be guided by IDIs conducted during Phase 1 and Phase 2. Our initial plan is to deliver MI-NAV in two waves. The first wave will be aimed at promoting uptake of PrEP at the prison, through the use of motivational interviewing. The second wave will be aimed at linking at-risk women to community-based PrEP care upon release from incarceration, by utilizing a patient navigator approach.
  Arms: MI-NAV
Behavioral: Standard of Care (SOC) — SOC will consist of a pamphlet regarding PrEP during incarceration, an offer of PrEP while incarcerated, and referral to community-based PrEP care upon release.
  Arms: Standard of Care (SOC)

SUMMARY:
Pre-exposure prophylaxis (PrEP) can be very effective at preventing HIV infection among women at high-risk for HIV but is underused in this population. Periods of incarceration represent an opportunity to identify women at risk and link them to PrEP care as they leave jail or prison. This study aims to improve linkage to community-based PrEP care to reduce HIV acquisition in a high-need, underserved community.

DETAILED DESCRIPTION:
Incarcerated women engage in high rates of sex- and drug-related behavior that place them at risk for HIV. Pre-exposure prophylaxis (PrEP) is an efficacious means of reducing HIV acquisition. There is a general lack of knowledge regarding PrEP among women at elevated risk, and only a small percentage of at-risk women are currently engaged in PrEP care. The period of incarceration represents an opportunity to identify at-risk women, initiate PrEP during incarceration, and establish linkage to community-based PrEP care upon release from incarceration. Further, post-release is a time period that is particularly risky, and there are numerous barriers that may impede linkage to community-based care in the absence of intervention.

To date, very little research has been done to improve linkage to PrEP care among US women. The proposed study will examine the acceptability, feasibility, and preliminary efficacy of a psychoeducation and motivational interviewing intervention to promote PrEP initiation during incarceration, followed by a patient navigator intervention to facilitate linkage to community-based PrEP care upon release from incarceration. The long-term goal of this line of research is to disseminate an efficacious PrEP Care linkage intervention for at-risk women post-release from incarceration. The present proposal seeks to develop intervention materials and conduct a small randomized controlled trial (RCT) of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth; at least 18 years of age; not currently pregnant; risk behavior prior to incarceration that meets CDC indications for PrEP; likely to be incarcerated for less than 6 months; able to understand and speak English and to provide written and verbal informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Rates of linkage to community-based PrEP care | 3 Months post-release
  Linkage to community-based care is operationalized as receipt of a prescription for PrEP from a community-based provider within 3 months of release from prison, confirmed through medical record data extraction.

SECONDARY OUTCOMES:
PrEP Adherence | 3 Months and 6 Months post-release
  PrEP adherence will be determined by drug concentrations in urine samples collected from participants who have been prescribed PrEP at 3 and 6 months. Presence of PrEP will be assessed with immunoassay developed by UrSure Inc.
PrEP Care Retention | 3 Month clinical appointments (+/- 1 month)
  PrEP retention in care will be defined as attending 3-month clinical appointments (+/- 1 month) which is in accordance with current CDC guidelines. This will be verified with medical records.
Alcohol and Drug Use | 6-months
  The Timeline Followback (TLFB) will be used to assess alcohol and drug use behavior at baseline, as well as during the follow-up interviews.
HIV Risk Behavior | 6-months
  The TLFB will be used to assess drug and sex risk behavior at baseline and during the follow-up interviews. In addition, the HIV Risk Assessment Battery will serve as a measure of overall sex and drug risk behavior.
Depressive Symptoms | 6-months
  The Center for Epidemiologic Studies Depression Scale (CES-D) will be administered at baseline and follow-up interviews to assess depressive symptoms
Treatment Received and Medications/Pregnancies | 6-months
  The Treatment Services Review (TSR) and Use of Medications Questionnaire will be used to measure the number and types of treatment services utilized, medications prescribed, and pregnancies experienced during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Ramsey SE, Ames EG, Brinkley-Rubinstein L, Teitelman AM, Clarke J, Kaplan C. Linking women experiencing incarceration to community-based HIV pre-exposure prophylaxis care: protocol of a pilot trial. Addict Sci Clin Pract. 2019 Mar 4;14(1):8. doi: 10.1186/s13722-019-0137-5. PMID 30832717